CLINICAL TRIAL: NCT07353372
Title: Interventional Study on Paraspinal Muscle Degeneration Leading to Lumbar Degenerative Diseases
Brief Title: Multimodal Exercise Therapy for Non-Surgical Intervention of Nonspecific Low Back Pain.
Acronym: METNLBP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: xuanwu_LBP
Record Dates: First submitted 2025-12-29; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Paraspinal Muscles; Low Back Pain; Machine Learning; Radiomics; Non-surgical Treatment
Keywords: Nonsteroidal anti-inflammatory drugs; Multidimensional exercise intervention
MeSH Terms: conditions — Low Back Pain | interventions — Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidimensional Exercise+Standard Oral Medication (Experimental): Participants receive a 6-week multidimensional exercise intervention (including aerobic, strength, balance, and flexibility training) combined with standard oral NSAIDs (e.g., ibuprofen or celecoxib) for 4 weeks
  Interventions: Behavioral: Multidimensional exercise intervention
- Standard Oral Medication Only (Active Comparator): Active ComparatorArm Description: Participants receive standard oral NSAIDs (e.g., ibuprofen or celecoxib) for 4 weeks without any structured exercise intervention.
  Interventions: Drug: Oral NSAIDs

INTERVENTIONS:
Behavioral: Multidimensional exercise intervention — Patients deemed by clinicians as not requiring surgical intervention and who consent to participate in the study will undergo an initial evaluation at the outpatient follow-up clinic. A multidimensional exercise intervention program and oral medication therapy (4 weeks) will be implemented based on the evaluation results.
  Arms: Multidimensional Exercise+Standard Oral Medication
Drug: Oral NSAIDs — Participants receive the same 4-week oral NSAID regimen without structured exercise intervention
  Arms: Standard Oral Medication Only

SUMMARY:
This multicenter, assessor-blinded, two-arm parallel randomized controlled trial (N = 314) will compare the efficacy and safety of a 6-week multidimensional exercise program plus usual pharmacological care (experimental arm) versus usual pharmacological care alone (control arm) in adults ≥ 60 years with chronic non-specific low-back pain (LBP) and imaging evidence of paraspinal muscle degeneration. The primary endpoint is change in Oswestry Disability Index (ODI) at 12 months. Secondary endpoints include pain VAS, JOA score, recurrence rate, and patient satisfaction measured repeatedly to 12 months. Advanced MRI radiomics and machine-learning algorithms will be used to build a "paraspinal muscle imaging-function-prognosis" prediction model and an open-access web tool for risk stratification. The study will generate a standardized, evidence-based non-operative care pathway for chronic LBP driven by paraspinal muscle degeneration

DETAILED DESCRIPTION:
Primary: to determine whether a 6-week supervised home-based multidimensional exercise program (aerobic, strength, balance, flexibility) added to short-term NSAIDs improves 12-month functional outcome (ODI) compared with NSAIDs alone.

Secondary: (1) compare pain intensity, quality of life, recurrence, and safety between arms; (2) develop and validate a radiomics-plus-machine-learning model that uses baseline MRI features of paraspinal muscles, demographic, clinical, and functional variables to predict treatment response and recurrence risk; (3) integrate the validated model with the exercise intervention to create a risk-stratified, early-intervention clinical pathway for chronic LBP.

Study Design：Multicenter, prospective, assessor-blinded, superiority RCT with 1:1 allocation, conducted at 4 tertiary hospitals and 1 academic research center in Beijing. Randomization (block sizes 4 and 6, stratified by center and sex) generated centrally via web-based system; allocation concealed from outcome assessors and statisticians.

Population Inclusion: age ≥ 60 y; LBP ≥ 3 months; ODI 20-60; MRI evidence of paraspinal muscle fatty infiltration ≥ Goutallier grade 2; no surgical indication; able to exercise.

Exclusion: specific spinal pathology (infection, tumor, fracture, severe deformity); previous lumbar surgery; severe comorbidities limiting exercise; cognitive impairment; current participation in another trial.

Interventions Experimental: 6-week multidimensional exercise (5 days/week, 30-40 min) plus 4-week oral NSAIDs (celecoxib or acetaminophen, dose-adjusted). Exercise comprises (1) low-intensity aerobic walking; (2) light-load high-repetition strength training (upper limb, lower limb, core); (3) balance and proprioceptive drills; (4) stretching. Printed manual + training diary; weekly phone/video supervision; compliance algorithm (≥ 75 % overall score required).

Control: same NSAID regimen alone. Both groups receive standardized education booklet on posture and activity pacing.

Outcomes Primary: ODI at 12 months (minimal clinically important difference 10 points). Secondary: VAS pain, JOA score at 1, 3, 6, 12 months; recurrence (≥ 24 h LBP with VAS > 2) within 12 months; patient satisfaction (NASS questionnaire); adverse events; compliance.

Imaging: axial MRI (3 T) at L1-5; semi-automated segmentation (3D-Slicer) to quantify cross-sectional area, fat fraction, radiomic features (shape, first-order, GLCM, GLRLM, GLSZM, GLDM).

Functional: Biering-Sørensen endurance test; surface electromyography of multifidus.

Biomarkers: baseline bloods (CBC, renal, hepatic panels). Sample Size 314 participants (157 per arm) provide 80 % power (α = 0.025 one-sided) to detect 15-point ODI difference (SD 15), allowing 10 % attrition.

Data Analysis

Intention-to-treat primary analysis: ANCOVA adjusted for baseline ODI, sex, center. Secondary longitudinal scores analyzed with mixed-effects models; recurrence with Kaplan-Meier and Cox regression.Radiomics:

7:3 split; 100× bootstrap; LASSO feature selection; multivariable modeling (logistic regression, random forest, XGBoost, LightGBM, MLP); performance reported as AUC, sensitivity, specificity, PPV, NPV, F1; SHAP/LIME for interpretability. Internal 5-fold cross-validation; final model deployed as web calculator.

Quality & Ethics Protocol approved by central ethics committee; registered at Chictr.org.cn. Written informed consent. Data entry via validated EpiData system; double verification; 5-year retention. Adverse events monitored by independent DSMB. Study conducted in accordance with Helsinki Declaration and ICH-GCP.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years
2. Chronic low-back pain for > 3 months (no surgical indication)
3. Planned to receive conservative treatment
4. Willing to participate and able to provide written informed consent

Exclusion Criteria:

1. Specific low-back pain due to infection, tumour, fracture, ankylosing spondylitis, scoliosis, or other structural spinal disorders
2. Previous lumbar surgery or current surgical indication for lumbar disease 3.Severe cardiopulmonary, hepatic or renal insufficiency that precludes exercise or drug therapy

4.Severe cognitive impairment or psychiatric disorder preventing cooperation 5.Marked exercise limitations or physical disability precluding rehabilitation training 6.Participation in another clinical trial that could interfere with outcomes 7.Known hypersensitivity to any study medication

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index(ODI) score at 1 year post-treatment | 12 months after randomization

SECONDARY OUTCOMES:
1.Change in Oswestry Disability Index (ODI) score. | Baseline, end-of-intervention, 1 month, 3 months, 6 months post-intervention
atient satisfaction with treatment(Assessed by the North American Spine Society (NASS) satisfaction questionnaire) | 12 months post-intervention
Change in Visual Analogue Scale (VAS) score for low back pain | Baseline, end-of-intervention, 1 month, 3 months, 6 months post-intervention
Change in Japanese Orthopaedic Association (JOA) score | Baseline, end-of-intervention, 1 month, 3 months, 6 months post-intervention
Recurrence rate of low back pain(Defined as new episode lasting ≥24 h with VAS) | Baseline, end-of-intervention, 1 month, 3 months, 6 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Shibao Lu, MD, Study Chair — Xuanwu Hospital, Beijing; Xiaolong Chen, MD, Study Director — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No